CLINICAL TRIAL: NCT06490328
Title: A Phase 3, Multi-center, Single-group, Open-label Study to Evaluate the Efficacy and Safety of DKF-MA102 in Patients With Prostate Cancer
Brief Title: Efficacy and Safety of DKF-MA102 in Patients With Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DKF-MA102-P3-1
Record Dates: First submitted 2024-06-13; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Advanced Prostate Cancer
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Intervention Model Description: Advanced Prostate Cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DKF-MA102 (Experimental): Leuprorelin acetate
  Interventions: Drug: DKF-MA102

INTERVENTIONS:
Drug: DKF-MA102 — Administered twice at 12-week intervals
  Other Names: Leuprorelin acetate

SUMMARY:
A phase 3, multi-center, single-group, open-label study to evaluate the efficacy and safety of DKF-MA102 in patients with prostate cancer.

DETAILED DESCRIPTION:
This study is conducted to confirm the pharmacodynamic effects, efficacy, and safety of DKF-MA102 in prostate cancer patients by measuring the changes in serum testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male aged 19 or older
2. Histologically or cytologically-confirmed prostate cancer
3. Serum testosterone level >150 ng/dL
4. ECOG PS grade ≤ 2
5. Life expectancy of at least 1 year

Exclusion Criteria:

1. History of surgical procedures such as testicular resection, adrenal resection, and pituitary resection
2. History of hormone therapy
3. History of 5α-reductase inhibitor
4. History of radical radiation therapy
5. History of adjuvant male hormone block therapy
6. Severe liver failure
7. Serum creatinine ≥1.5 times the ULN
8. Hormone-independent prostate cancer
9. Diagnosed pituitary adenoma
10. Brain metastasis or spinal cord compression
11. Requires prostatectomy, radiation therapy, chemotherapy, and anti-androgen therapy during the clinical trial period
12. Urinary tract obstruction
13. Cardiovascular disease
14. Significant impairments in the digestive system, respiratory system, endocrine system, and central nervous system
15. Uncontrolled diabetes
16. Allergic reaction or hypersensitivity to any ingredient of the investigational product or to a synthetic GnRH or GnRH analogs
17. Severe asthma, severe vascular edema, and severe hives
18. Significant infection
19. Lack of self-determination due to psychiatric illness
20. Participating in another interventional clinical trial
21. Pregnant or unwilling to use medically approved contraception
22. Deemed inappropriate to participate in this clinical trial by the investigator

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants | Week 4
  Percentage of participants with testosterone suppression(≤ 50ng/dL) at Week 4
Percentage of participants | Week 24
  Percentage of participants with testosterone suppression(≤ 50ng/dL) from Week 4 to Week 24

SECONDARY OUTCOMES:
Serum luteinizing hormone(LH) levels | Week 24
  Changes in serum luteinizing hormone(LH) levels from baseline to Weeks 4, 12 and 24
Serum prostate specific antigens(PSA) | Week 24
  Changes in serum prostate specific antigens(PSA) from baseline to Weeks 4, 12 and 24
Percentage of participants | Week 24
  Percentage of participants with testosterone suppression(≤ 20ng/dL) from Week 4 to Week 24
Quality of life(FACT-P) | Week 24
  Comparative evaluation of quality of life(FACT-P) of subjects from baseline to Weeks 4, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Choung-Soo Kim, M.D.,Ph.D, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University mokdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No